CLINICAL TRIAL: NCT02967289
Title: A Phase III, Randomised, International Trial Comparing mFOLFIRINOX Triplet Chemotherapy to mFOLFOX for High-risk Stage III Colon Cancer in Adjuvant Setting
Brief Title: IRinotecan and Oxaliplatin for Colon Cancer in Adjuvant Setting
Acronym: IROCAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Canadian Cancer Trials Group (Network); GONO GROUP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0110/1609_PRODIGE52/UCGI29; 2016-001491-29 (EudraCT Number)
Record Dates: First submitted 2016-11-09; First posted 2016-11-18 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer (High-risk Stage III: pT4N1 or pT1 to 4 N2)
Keywords: colon; cancer; stage 3; high-risk; mFolfirinox; mFolfox6; adjuvant
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms | interventions — Irinotecan; Folfox protocol; Leucovorin; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: The trial is a phase III, multicenter, open-labeled randomized trial comparing the association 5-fluorouracil, folinic acid, irinotecan and oxaliplatin (mFOLFIRINOX) versus oxaliplatin, folinic acid, 5FU (mFOLFOX 6) chemotherapy protocols in patients with high-risk stage III colon cancer in the adjuvant setting.
Masking Description: The primary end-point is the Disease Free Survival (DFS) at 3 years, defined as the time from the date of randomization up to the date of:
  * first local, regional or distant relapse;
  * second colorectal cancer;
  * death from any cause included treatment-related death. Other primary cancer (except second primary colorectal) will be ignored. Second primary cancer will be recorded to have the opportunity of evaluating other definition of DFS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): mFOLFIRINOX Folfox Protocol + Irinotecan
  Interventions: Drug: Irinotecan; Drug: Folfox Protocol
- Arm B (Active Comparator): mFOLFOX 6 Folfox Protocol
  Interventions: Drug: Folfox Protocol

INTERVENTIONS:
Drug: Irinotecan — every 14 days, 12 cycles, 24 weeks, new cycle beginning on day 15: irinotecan (Campto®) 180 mg/m² on D1, IV infusion over 90 minutes to begin 30 min after folinic acid infusion is started
  Other Names: Campto
  Arms: Arm A
Drug: Folfox Protocol — every 14 days, 12 cycles, 24 weeks, new cycle beginning on day 15: oxaliplatin (Eloxatin®) 85 mg/m² on D1, IV infusion over 2 hours, followed by folinic acid 400 mg/m² (racemic mixture) (or 200 mg/m² if L-folinic acid) IV infusion over 2 hours 5-FU 2400 mg/m²/h IV continuous infusion over 46 hours starting at the end of folinic acid infusion
  Other Names: acid folinic + oxaliplatine + 5-FU

SUMMARY:
The trial is a phase III, multicenter, open-labeled randomized trial comparing the association of 5-fluorouracil (5-FU), folinic acid, irinotecan, and oxaliplatin (mFOLFIRINOX) versus oxaliplatin, folinic acid, and 5-FU (mFOLFOX 6) chemotherapy protocols in patients with high-risk stage III colon cancer in the adjuvant setting.

DETAILED DESCRIPTION:
After inclusion and non-inclusion criteria have been fulfilled and the patient consent has been obtained, the patient will be included and randomized in the trial. The maximum delay allowed between the signature of the consent form by the patient and the randomization in the study is 28 days.

The randomization procedure using minimization method will allocate the treatments mFOLFIRINOX or mFOLFOX 6 with a 1:1 ratio, and will be stratified by the following criteria:

* Perforation or urgent surgery versus no perforation and no urgent surgery.
* T1-T3N2 vs T4aN1 versus T4bN1 versus T4N2.
* Right colon (right of splenic flexure) vs left colon.
* Country (France vs Canada vs Italy). Patient eligible and who have signed the informed consent will be randomized in one of the two treatments arms and will receive every 14 days their treatment for a duration of 12 cycles.

Arm A: mFOLFIRINOX Arm B: mFOLFOX 6

ELIGIBILITY:
DIAGNOSIS AND INCLUSION CRITERIA:

1. Patient ≥18 years and < 75 years
2. Patient ≥18 years and <71 years must have an ECOG ≤1 - Patients ≥71 years and < 75 years must have an ECOG = 0
3. Pathologically confirmed high-risk stage III colon adenocarcinoma, restricted to pT4N1 or pT1-4N2 tumor.
4. Curative R0 surgical resection.
5. Patients who have undergone surgery for colon cancer, defined as a tumor location >12 cm from the anal verge by endoscopy and/or above the peritoneal reflection at surgery (high rectum), without gross or microscopic evidence of residual disease after surgery with curative intent
6. Start of study drug treatment has to be performed less than 56 days after surgery.
7. No prior chemotherapy.
8. No prior abdominal or pelvic irradiation.
9. Patient with adequate organ function:

   * Absolute neutrophil count (ANC) ≥ 2 x 109/L
   * Haemoglobin ≥9 g/dL
   * Platelets (PTL) ≥100 x 109/L
   * AST/ALT ≤2.5 x ULN
   * Alkaline phosphatase ≤2.5 x ULN
   * Total Bilirubin ≤1.5 x ULN (Upper Limit of Normal)
   * Creatinine clearance ≥50 mL/min (Cockcroft and Gault formula)
   * Kalemia, magnesemia, calcemia ≥ 1 LLN (Lower Limit of Normal)
   * Carcinoembryonic antigen (CEA) ≤10ng/mL after surgery (during screening period)
10. Adequate contraception if applicable.
11. Patient able and willing to comply with study procedures as per protocol
12. Patient able to understand and willing to sign and date the written voluntary informed consent form at screening visit prior to any protocol-specific procedures
13. Public or private health insurance coverage
14. Life expectancy of > or = at 5 years
15. Uracilemia < 16 ng/ml (only for french centers)

Exclusion Criteria:

1. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to study treatment start. Incompletely healed wounds or anticipation of the need for major surgical procedure during the course of the study
2. Metastatic disease
3. Presence of inflammatory bowel disease and/or ileus
4. Known hypersensitivity reaction to any of the components of study treatments.
5. Pregnancy (absence to be confirmed by β-hCG test) or breast-feeding period
6. Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia (for men: QTc ≥450 msec, for women: QTc ≥470 msec)
7. Previous malignancy in the last 5 years except curative treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
8. Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
9. History or current evidence on physical examination of central nervous system disease or peripheral neuropathy ≥ grade 1 Common Toxicity Criteria for Adverse Events (CTCAE) v4.03.
10. Any significant disease which, in the investigator's opinion, would exclude the patient from the study.
11. Patient with a DPD deficiency or UGT1A1 homozygous 7/7; the test should be done for all patients before 5-FU administration, according to ANSM communication regarding recommendation about high risk of no testing DPD in patient before 5-FU administration; (Appendices 8 to 11).
12. Patients already included in another therapeutic trial involving an experimental drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 YEARS after inclusion
  DFS :
  defined as the time from the date of randomization up to the date of:
  * first local, regional or distant relapse;
  * second colorectal cancer;
  * death from any cause included treatment-related death.

SECONDARY OUTCOMES:
Disease Free Survival | 2 YEARS after inclusion
  DFS :
  defined as the time from the date of randomization up to the date of:
  * first local, regional or distant relapse;
  * second colorectal cancer;
  * death from any cause included treatment-related death.
Overall Survival | 5 YEARS after inclusion
  Overall Survival (OS) is defined as the time from the date of randomization to the date of documented death from any cause
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 YEARS after inclusion
  Safety of the study treatment will be assessed on occurrence of Adverse Events (AEs), intake of concomitant treatments, per-treatment arising changes in physical examination, vital signs (blood pressure, pulse rate and body temperature), ECG, and clinical laboratory tests (biochemistry, haematology). Safety parameters will be graded based on NCI CTCAE v4.03 classification.
  The following parameters will be particularly followed:
  The incidence of haematological toxicities (grade 3-4, in particular neutropenia and febrile neutropenia); The incidence of GI toxicities, in particular diarrhea; The incidence of peripheral neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, Professor, Study Chair — Hôpital FOCH, SURESNES; Julien TAIEB, Professor, Study Chair — Hôpital Européen Georges-Pompidou, PARIS; Thierry ANDRE, Professor, Study Chair — AP-HP Hôpital Saint-Antoine, PARIS
Locations (17):
- Canada (4):
  - The PEI Cancer Treatment Centre Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- France (13):
  - Institut de Cancérologie de l'Ouest -site Paul Papin, Angers
  - CHD de Vendée, La Roche-sur-Yon
  - Ch Emile Roux, Le Puy-en-Velay
  - Hospices civils de Lyon - Hôpital Edouard Herriot, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Icm Val D'Aurelle, Montpellier
  - Institut de Cancérologie de l'Ouest -site René Gauducheau, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Annecy Genevois, Pringy
  - Institut Jean Godinot, Reims
  - CHP Saint Grégoire, Saint-Grégoire
  - Clinique de la Côte d'Emeraude, St-Malo

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Bennouna J, Andre T, Campion L, Hiret S, Miglianico L, Mineur L, Touchefeu Y, Artru P, Asmis T, Bouche O, Borde F, Kavan P, Lam YH, Rajpar LS, Emile JF, Jouffroy C, Gill S, Taieb J. Rationale and Design of the IROCAS Study: Multicenter, International, Randomized Phase 3 Trial Comparing Adjuvant Modified (m) FOLFIRINOX to mFOLFOX6 in Patients With High-Risk Stage III (pT4 and/or N2) Colon Cancer-A UNICANCER GI-PRODIGE Trial. Clin Colorectal Cancer. 2019 Mar;18(1):e69-e73. doi: 10.1016/j.clcc.2018.09.011. Epub 2018 Oct 19. PMID 30415988